CLINICAL TRIAL: NCT01618591
Title: A Randomized, Double-Blind, Clinical Trial Evaluating Three Single Dose Regimens With Loperamide for Treatment of Ambulatory Watery Travelers' Diarrhea, and Azithromycin With and Without Loperamide for Treatment of Ambulatory Dysentery/Febrile Diarrhea
Brief Title: Trial Evaluating Ambulatory Treatment of Travelers' Diarrhea
Acronym: TrEAT TD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: AWD arm was completed. ADF diarrhea arm was unable to fill completely and there are no funds remaining to continue recruiting/enrolling.
Sponsor: Uniformed Services University of the Health Sciences (U.S. Federal Agency)
Collaborators: Navy Bureau of Medicine and Surgery (U.S. Federal Agency); Ministry of Defence, United Kingdom (Other Government); Naval Medical Research Center (U.S. Federal Agency); Naval Medical Research Unit- 3 (U.S. Federal Agency); United States Army Medical Unit - Kenya (U.S. Federal Agency); United States Naval Medical Center, Portsmouth (U.S. Federal Agency); Naval Medical Research Unit- 6 (U.S. Federal Agency)
Responsible Party: Principal Investigator, Mark Riddle, CDR, MC, USN, Head, Enteric Diseases Department, Naval Medical Research Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IDCRP-065
Record Dates: First submitted 2012-06-01; First posted 2012-06-13 (Estimated); Last update posted 2016-11-28 (Estimated); Status verified 2016-11

CONDITIONS: Acute Watery Diarrhea; Dysentery/Febrile Diarrhea
Keywords: diarrhea; travelers' diarrhea; watery diarrhea; enteric illness; dysentery; gastrointestinal
MeSH Terms: conditions — Dysentery; Diarrhea | interventions — Rifaximin; Azithromycin; Levofloxacin; Loperamide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Acute Watery Diarrhea (Experimental)
  Interventions: Drug: Single dose rifaximin 1650 mg; Drug: Single dose azithromycin 500 mg; Drug: Single dose levofloxacin 500 mg
- Acute Dysentery/Febrile (Experimental)
  Interventions: Drug: Single dose azithromycin 1000 mg plus loperamide; Drug: Single dose azithromycin 1000 mg plus placebo

INTERVENTIONS:
Drug: Single dose rifaximin 1650 mg — Rifaximin 1650 mg as a single dose plus loperamide 4 mg initially followed by 2 mg after each unformed stool, not to exceed 16 mg/day for 2 days
  Arms: Acute Watery Diarrhea
Drug: Single dose azithromycin 500 mg — Azithromycin 500 mg as a single dose plus loperamide 4 mg initially followed by 2 mg after each unformed stool, not to exceed 16 mg/day for 2 days
  Arms: Acute Watery Diarrhea
Drug: Single dose levofloxacin 500 mg — Levofloxacin 500 mg as a single dose plus loperamide 4 mg initially followed by 2 mg after each unformed stool, not to exceed 16 mg/day for 2 days
  Arms: Acute Watery Diarrhea
Drug: Single dose azithromycin 1000 mg plus loperamide — Azithromycin 1000 mg as a single dose plus loperamide 4 mg initially followed by 2 mg after each unformed stool, not to exceed 16 mg/day for 2 days
  Arms: Acute Dysentery/Febrile
Drug: Single dose azithromycin 1000 mg plus placebo — Azithromycin 1000 mg as a single dose and placebo in lieu of loperamide
  Arms: Acute Dysentery/Febrile

SUMMARY:
The purpose of the trial is to develop the evidence on relative efficacy of 3 available single-dose loperamide adjuncted regimens for watery diarrhea and a single-dose regimen, with and without loperamide, for dysentery/febrile diarrhea required for informing decisions among these regimens. Information from this study will be used to develop management guidelines for the diagnosis and management of travelers' diarrhea (TD) among deployed United States and United Kingdom military personnel.

DETAILED DESCRIPTION:
The study will be a multi-site, randomized, double-blind, controlled clinical trial among ambulatory deployed personnel. Patients presenting for care will be clinically assessed and a determination made as to whether they have acute watery diarrhea (AWD) or acute dysentery/febrile diarrhea (ADF). For the AWD arm, patients will be randomized to receive 1 of 3 regimens: (1) rifaximin 1650 mg as a single dose plus loperamide 4 mg initially followed by 2 mg after each unformed stool, not to exceed 16 mg/day for 2 days (120 subjects); (2) azithromycin 500 mg as a single dose plus loperamide 4 mg initially followed by 2 mg after each unformed stool, not to exceed 16 mg/day for 2 days (120 subjects); or (3) levofloxacin 500 mg as a single dose plus loperamide 4 mg initially followed by 2 mg after each unformed stool, not to exceed 16 mg/day for 2 days (120 subjects).

For the ADF arm, patients will be randomized to receive 1 of 2 regimens: (1) azithromycin 1000 mg as a single dose plus loperamide 4 mg initially followed by 2 mg after each unformed stool, not to exceed 16 mg/day for 2 days (75 subjects); or (2) azithromycin 1000 mg as a single dose without loperamide (75 subjects).

Study Procedures (Brief): Baseline exam as well as blood and stool samples will be collected at initial clinic visit. Clinical assessments will be performed at 24 hours, 72 hours, and 7 days. In addition, microbiological cure will be evaluated at 7-d post initiation of treatment. Subjects will have blood drawn to assess for serological conversion to common enteric pathogens, and stool collected at 7- and 21-d . Subjects may also opt in for long-term follow-up at time of enrollment, which will assess for development of post-infectious functional bowel disorders. All subjects will complete a baseline assessment at 7-d visit, and those who opt for the additional follow-up will complete a series of web-based surveys at 3-, 6-, 9-, and 12-m post enrollment.

ELIGIBILITY:
Inclusion Criteria:

1. Active duty military or military beneficiary, 18 years-old or older.
2. Presence of acute diarrhea (3 or more stools in 24 hours or 2 or more stools in 24 hours and associated symptoms such as nausea, vomiting, abdominal cramps or tenesmus) and <96 hours duration.
3. Eligible for ambulatory management.
4. Able to comply with follow-up procedures.
5. Will remain in country for at least 7 days

Exclusion Criteria:

1. Allergy to rifamycins, quinolones, macrolides, or loperamide (not including mild gastrointestinal upset).
2. Antibiotic therapy in the 72 hours prior to presentation (excluding malaria prophylaxis with mefloquine, malarone, chloroquine/proguanil, or doxycycline).
3. Concomitant medications with known drug-drug interactions with any of the study drugs (includes theophylline, digoxin, and warfarin).
4. History of seizures (relative contraindication to quinolones)
5. Positive pregnancy test at presentation (contraindicated with fluoroquinolone therapy). All female subjects will be administered a urine pregnancy test prior to enrollment.
6. Presence of symptoms >96 hours prior to initiating treatment.
7. Use of >4 mg loperamide or use of any amount of loperamide for greater than 24 hours prior to enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 384 (Actual)
Dates: Start 2012-09; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Clinical Cure - Acute Watery Diarrhea group | 24 hours
  * No grade 3-5 stools beyond 24 hours after initiation of therapy meeting diarrhea definition (≥3 loose or liquid stools in 24 hour period). All diarrhea associated symptoms present must be no greater than mild in severity and have no impact on activity.
  * AND, no treatment failure events to include the following:
    * Recurrence of diarrheal illness meeting case definition of TD occurring within 72 hours after clinical cure
    * Worsening of, or failure to improve, clinical symptoms after 24 hours of therapy
    * Illness continuing after 72 hours
Clinical Cure - Acute Dysentery/Febrile Diarrhea group | 48 hours
  * No grade 3-5 stools beyond 48 hours after initiation of therapy meeting diarrhea definition (≥3 loose or liquid stools in 24 hour period) and resolution of acute dysentery/febrile diarrhea-associated signs/symptoms to include fever and gross blood in stool, as well as report of no impact on activity
  * AND, no treatment failure events to include the following:
    * Recurrence of diarrheal illness meeting case definition of TD occurring within 72 hours after clinical cure
    * Worsening of, or failure to improve after 24 hours of therapy
    * Illness continuing after 72 hours

SECONDARY OUTCOMES:
Time to Last Unformed Stool | 24, 48, 72 hours
  Calculated as the time from taking the first dose of study medication until passage of the last unformed stool that meets diarrhea definition (grade 3-5 stool associated with 2 other loose stools in 24 hours or 1 other loose stool and associated symptoms in that same 24 hour block) after which subjects are declared well. Where, last unformed stool = last grade 3-5 stool occurring in a 24-hr period meeting the diarrhea definition.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Riddle, MD, DrPH, Principal Investigator — Naval Medical Research Center
Locations (5):
- UK Role 3 Joint Force Hospital, Camp Bastion Air Base, Afghanistan
- U.S. Naval Expeditionary Base, Camp Lemonnier, Djibouti
- Joint Task Force - Bravo, Soto Cano Air Base, Honduras
- British Army Training Unit Kenya, Nanyuki, Kenya
- Armed Forces Research Institute of Medical Sciences, Bangkok, Thailand

REFERENCES:
- [Derived] Johnson RC, Van Nostrand JD, Tisdale M, Swierczewski B, Simons MP, Connor P, Fraser J, Melton-Celsa AR, Tribble DR, Riddle MS. Fecal Microbiota Functional Gene Effects Related to Single-Dose Antibiotic Treatment of Travelers' Diarrhea. Open Forum Infect Dis. 2021 May 28;8(6):ofab271. doi: 10.1093/ofid/ofab271. eCollection 2021 Jun. PMID 34189178
- [Derived] Riddle MS, Connor P, Fraser J, Porter CK, Swierczewski B, Hutley EJ, Danboise B, Simons MP, Hulseberg C, Lalani T, Gutierrez RL, Tribble DR; TrEAT TD Study Team. Trial Evaluating Ambulatory Therapy of Travelers' Diarrhea (TrEAT TD) Study: A Randomized Controlled Trial Comparing 3 Single-Dose Antibiotic Regimens With Loperamide. Clin Infect Dis. 2017 Nov 29;65(12):2008-2017. doi: 10.1093/cid/cix693. PMID 29029033